CLINICAL TRIAL: NCT02974530
Title: Description and Modeling of Swallowing Disorders After a Stroke
Acronym: AVC-MODE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: National Research Agency, France (Other); University Hospital, Caen (Other); University Hospital, Montpellier (Other); Centre Hospitalier du Pays d'Aix (Other); Université Joseph Fourier (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A00070-51
Record Dates: First submitted 2016-09-01; First posted 2016-11-28 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2016-08

CONDITIONS: Stroke; Swallowing Disorders
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Magnetic Resonance Spectroscopy; Voice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stroke population: Patient with stroke will be explored during their acute phase and in 6 months of diagnosis.
  Interventions: Other: Neurological evaluation; Other: Laryngological evaluation; Other: MRI evaluation; Other: Breathing investigation; Other: Postural investigation; Other: Voice and soundscape investigation
- Healthy population: Healthy subjects will be explored in Grenoble in research laboratory
  Interventions: Other: Breathing investigation; Other: MRI and articulatory investigation; Other: Postural investigation; Other: Voice and soundscape investigation

INTERVENTIONS:
Other: Neurological evaluation
  Groups: Stroke population
Other: Laryngological evaluation
  Groups: Stroke population
Other: MRI evaluation
  Groups: Stroke population
Other: Breathing investigation
Other: MRI and articulatory investigation
  Groups: Healthy population
Other: Postural investigation
Other: Voice and soundscape investigation

SUMMARY:
The oropharyngeal junction participates in 3 interpenetrating functions: Swallowing, Breathing and Speech. In the context of ischemic or hemorrhagic stroke, these are altered, isolated or associated manner, causing major disorders and representing a source of handicap for patients.

Understanding the swallowing mechanisms is therefore a major challenge to guide the rehabilitation and improve the initial and long-term prognosis of patients with stroke.

The main objective of this study is to describe and modeling, thanks to a clinical, physiological and radiological knowledge base, swallowing, speech and breathing, in patients with stroke and in healthy subjects.

ELIGIBILITY:
For patients after stroke

Inclusion Criteria:

* First stroke confirmed by MRI < 15 days
* No severe leukoaraiosis
* Swallowing disorders identified (GUSS scale < 20)
* Neurological deficit identified (NIHSS scale <15)
* Patient able to cooperate for investigations
* Informed consent signed

Exclusion Criteria:

* Cerebral hemorrhage
* History of neurological disease that can lead to swallowing disorders
* History of laryngological disease such as previous surgery or radiation neck
* Tracheotomy
* Vigilance disorders
* Pregnant, parturient or nursing woman
* Protected adult
* Simultaneous participation in another study
* Non registered to the French social security system

For healthy subjects

Inclusion Criteria :

* Age between 18 and 40 years old
* French native speaker
* Normal hearing with or without corrective
* No oral or written language disorders
* No neurological or psychiatric disorders
* Informed consent signed

Exclusion Criteria

* MRI contraindication
* Pregnant, parturient or nursing woman
* Simultaneous participation in another study
* Non registered to the French social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Multicenter study with two cohorts unpaired : first of healthy subjects / second of patient with ischemic stroke.
  Study size expected :
  * 120 stroke patients in 4 University Hospital
  * 30 healthy subjects explored in research laboratory
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change of Clinical severity score | At inclusion and 6 months after diagnosis
  NIHSS scale
Change of swallowing disorder | Within 15 days after diagnosis and 6 months after diagnosis
  Test : GUgging Swallowing Screen

SECONDARY OUTCOMES:
Change of aphasia disorder | Within 15 days after diagnosis and 6 months after diagnosis
  Questionnaire : Aphasia rapid test
Change of state of depression and anxiety | Within 15 days after diagnosis and 6 months after diagnosis
  Questionnaire : anxiety and depression scale
Change of behavioural attention | Within 15 days after diagnosis and 6 months after diagnosis
  Questionnaire : Catherine Bergego scale

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hospital, Aix-en-Provence
  - University hospital, Caen
  - University hospital, Grenoble
  - University hospital, Montpellier

IPD SHARING:
Plan to Share IPD: No